CLINICAL TRIAL: NCT00000854
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I/II Trial of Nandrolone Decanoate in Women With HIV-Associated Weight Loss
Brief Title: A Study to Evaluate the Effect of Nandrolone Decanoate in Women With HIV-Associated Weight Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 329; 11301 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Placebos; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Anabolic Steroids; HIV Wasting Syndrome; nandrolone decanoate
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nandrolone Decanoate

INTERVENTIONS:
Drug: Nandrolone decanoate

SUMMARY:
The purpose of this study is to see if giving nandrolone decanoate (a hormonal drug) will cause weight gain in HIV-positive women who have HIV-associated weight loss (wasting).

Wasting has become an AIDS-defining condition. In the past, most studies that examined wasting treatments were limited to men. However, it appears that wasting in HIV-positive men is linked to levels of testosterone (a hormone which affects men's bodies more than women's). This study has been designed for women only, in order to best treat wasting in HIV-positive women.

DETAILED DESCRIPTION:
Body wasting is an increasingly frequent AIDS-defining condition and it is becoming evident that women are not exempt from this complication of HIV. Although multicenter trials of megestrol acetate, dronabinol and growth hormone have not specifically excluded women, women have generally been underrepresented in these trials. This study hopes to generate data that will be substantial enough to perform an analysis that might determine whether there are gender-based differences in anabolic potential.

Patients will be randomized to receive either nandrolone decanoate or placebo every 2 weeks for 12 weeks of the study. All patients who complete the first 12 weeks of the study will be eligible to receive open-label nandrolone for the subsequent 12 weeks.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are an HIV-positive woman over 13 years old (need consent if under 18).
* Have lost weight over the past 12 months.
* Are able to eat almost enough to maintain your current weight.
* Agree to practice abstinence or use effective methods of birth control.
* Are on a stable anti-HIV drug regimen or have not been on any anti-HIV drug regimen for the past 30 days.

Exclusion Criteria

You will not be eligible for this study if you:

* Are allergic to nandrolone.
* Have a history of cervical cancer, diabetes, cardiomyopathy or congestive heart failure, or are taking certain medications.
* Have an active opportunistic (HIV-associated) infection or another major illness within 30 days of study entry.
* Have an abnormal PAP smear.
* Have difficulty eating (are on tube-feeding, for example).
* Have severe nausea, vomiting, or diarrhea.
* Have Kaposi's sarcoma (unless stable) or are receiving chemotherapy or radiation for any type of cancer.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Mulligan, Study Chair; R Clark, Study Chair; J Currier, Study Chair
Locations (22):
- United States (20):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
- Puerto Rico (2):
  - Puerto Rico-AIDS CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Mulligan K, Zackin R, Clark RA, Alston-Smith B, Liu T, Sattler FR, Delvers TB, Currier JS; AIDS Clinical Trials Group 329 Study Team; National Institute of Allergy and Infectious Diseases Adult AIDS Clinical Trials Group. Effect of nandrolone decanoate therapy on weight and lean body mass in HIV-infected women with weight loss: a randomized, double-blind, placebo-controlled, multicenter trial. Arch Intern Med. 2005 Mar 14;165(5):578-85. doi: 10.1001/archinte.165.5.578. PMID 15767536